CLINICAL TRIAL: NCT01871519
Title: A Prospective and Multicenter Evaluation of Outcomes for Quality of Life and Activities of Daily Living for Balloon Kyphoplasty in the Treatment of Vertebral Compression Fractures
Brief Title: Evaluation of Outcomes for Quality of Life and Activities of Daily Living for BKP in the Treatment of VCFs
Acronym: EVOLVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P12-03
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Compression Fracture of Vertebral Body; Osteoporosis; Cancer
Keywords: vertebral body compression fracture
MeSH Terms: conditions — Osteoporosis; Neoplasms | interventions — Kyphoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon Kyphoplasty (Other): This group of patients will be treated with balloon kyphoplasty in the treatment of painful, acute VCFs associated with either osteoporosis or cancer.
  Interventions: Device: Balloon kyphoplasty

INTERVENTIONS:
Device: Balloon kyphoplasty — The devices to be used in this study are intended for percutaneous balloon kyphoplasty (BKP) and consist of the Kyphon® bone access needles and cannulae, inflatable bone tamps, curettes, polymethyl methacrylate bone cement (PMMA) bone cements, and bone filler devices.
  Other Names: BKP

SUMMARY:
The study objective is to collect and report 12-month outcomes pertaining to activities of daily living, quality of life, and safety parameters in a Medicare population to be treated with balloon kyphoplasty in the treatment of painful, acute, vertebral body compression fractures (VCFs) associated with either osteoporosis or cancer. The primary objective is to show statistically significant improvement from baseline in the four co-primary endpoints (SF-36v2, PCS, EQ-5D, NRS back pain and ODI) at 3-months; study success will be declared if the primary objective is met. New radiographic fractures, non-surgical management received, VCF-related healthcare resource utilization, and vertebral body height restoration data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Identified as an appropriate candidate for BKP and should have made the choice to have the procedure.
2. Must be Medicare Eligible (At least 65 years of age or otherwise eligible).
3. Must have one to three target VCFs, located between T5 and L5, which are due to underlying primary or secondary osteoporosis or cancer.
4. Cancer patients should not have had a change in chemotherapy regimen within the last month, nor should they have a planned change within the next month from time of enrollment, with the exception of changes in dose.
5. All VCFs to be treated must have clinical pain symptoms (pain on palpation/percussion over the fractured vertebral body) that correlate with radiographic findings as follows:

   1. Height change: An acute (≤ four month) change in VB height or morphology from a previous x-ray, CT or MRI, with height loss at the anterior, middle or posterior portion of the VB consistent with a worsening of one or more grades by the Genant criteria20, OR
   2. Positive MRI or bone scan: VB shows hyperintense signal on STIR sequence MRI, or target VB is positive on radionuclide bone scan.
6. All VCFs to be treated must have an estimated fracture age of four months or less.
7. Treatment of all target VCFs must be technically feasible and clinically appropriate for balloon kyphoplasty.
8. Pre-treatment back pain by numerical rating scale (NRS) score must be ≥ 7 (0-10 scale) and refractory to non-surgical management.
9. Pre-treatment Oswestry Disability Index must be ≥30 (0 - 100 scale).
10. Must have life expectancy of ≥ 12 months.
11. Must declare availability for all study visits.
12. Must be able to understand the risks and benefits of participating in the study and be willing to provide written informed consent.
13. Must have the mental capacity necessary to comply with protocol requirements for the 12- month duration of study.

Exclusion Criteria:

1. Vertebral body morphology or fracture configuration contraindicative of balloon kyphoplasty.
2. VCFs due to high-energy trauma.
3. Asymptomatic VCFs or prophylactic treatment of non-fractured vertebral bodies.
4. VCFs accompanied at the same site by primary tumors of the bone (e.g., osteosarcoma), solitary plasmacytoma or osteoblastic tumors.
5. Platelet count of <20,000/uL as measured at the time of hospital admission for the procedure.
6. Back pain due to causes other than acute fracture.
7. VCF with a clinically estimated (based on radiographic evidence as well as patient history) age of fracture > four months.
8. VCF accompanied by objective evidence of secondary radiculopathy or neurologic compromise.
9. VCFs with the need for spinal surgery beyond balloon kyphoplasty.
10. Spinal cord compression or canal compromise requiring decompression.
11. Significant clinical comorbidity that may either contra-indicate surgery or interfere with long-term data collection or follow-up.
12. Pre-existing conditions contrary to balloon kyphoplasty such as:

    1. Allergy to any components (e.g., bone cement, contrast medium) of the balloon kyphoplasty device/procedure.
    2. Active or incompletely treated infection of the vertebral column or active systemic infection, including unresolved urinary tract infection.
    3. Irreversible coagulopathy or bleeding disorder.
13. Contraindications to both MRI and radionuclide bone scan.
14. Concurrent participation in another clinical study.
15. Pregnant or intending to become pregnant during the course of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 354 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham, Division of Neurological Surgery, Birmingham, Alabama
  - Washington Radiologist Medical Group, Fremont, California
  - Sutter Health Sacramento Sierra Region, Sacramento, California
  - Alta Orthopaedic Medical Group, Santa Barbara, California
  - Torrance Memorial Medical Center, Torrance, California
  - Radiology Imaging Specialist of Lakeland, Lakeland, Florida
  - The Back Center, Melbourne, Florida
  - Physicians & Surgeons of Pocatello, Blackfoot, Idaho
  - St. Luke's Health System, Boise, Idaho
  - Central Illinois Neuroscience Foundation, Bloomington, Illinois
  - Adventist Health Partners, Hinsdale, Illinois
  - Presence Saint Joseph Medical Center, Joliet, Illinois
  - Illinois Bone & Joint, Morton Grove, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Advanced Diagnostic Imaging, PC, Saginaw, Michigan
  - Beaumont Health System, Troy, Michigan
  - Premier Radiology, Tupelo, Mississippi
  - Sierra Regional Spine Institute, Reno, Nevada
  - Consulting Orthopaedic Associates, Inc, Sylvania, Ohio
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - James R. Webb, P.C., Tulsa, Oklahoma
  - NeuroSpine Institute, LLC, Eugene, Oregon
  - Scoliosis & Spine Surgery Clinic of Memphis, PLLC, Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee

REFERENCES:
- [Derived] Beall DP, Chambers MR, Thomas S, Amburgy J, Webb JR Jr, Goodman BS, Datta DK, Easton RW, Linville D 2nd, Talati S, Tillman JB. Prospective and Multicenter Evaluation of Outcomes for Quality of Life and Activities of Daily Living for Balloon Kyphoplasty in the Treatment of Vertebral Compression Fractures: The EVOLVE Trial. Neurosurgery. 2019 Jan 1;84(1):169-178. doi: 10.1093/neuros/nyy017. PMID 29547939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 354 subjects were enrolled in this study. Among them, 350 subjects had BKP surgery and 4 subjects were not treated with BKP. Two of the non-treated subjects voluntarily withdrew from the study and 2 subjects were lost-to-follow-up before surgery.
Groups:
- Balloon Kyphoplasty: This group of patients were treated with balloon kyphoplasty in the treatment of painful, acute VCFs associated with either osteoporosis or cancer.
  Balloon kyphoplasty: The devices to be used in this study are intended for percutaneous balloon kyphoplasty (BKP) and consist of the Kyphon® bone access needles and cannulae, inflatable bone tamps, curettes, polymethyl methacrylate bone cement (PMMA) bone cements, and bone filler devices.
Period: Overall Study
Arm/Group | Balloon Kyphoplasty
Started | 350
Completed | 260
Not Completed | 90
Not completed — Death | 26
Not completed — Lost to Follow-up | 15
Not completed — Withdrawal by Subject | 49

BASELINE CHARACTERISTICS:
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 344
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 12
  Black or African American | 4
  Native Hawaiian or other pacific islander | 0
  White | 330
  Other | 3
Height [Mean (Standard Deviation); unit: inches] | 64.3 (3.9)
Weight [Mean (Standard Deviation); unit: lbs] | 153.9 (36.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (5.5)
Estimated pre-fracture vertebral body height [Mean (Standard Deviation); unit: mm] — Population: A total of 490 treated levels in 344 subjects were included in vertebral body height restoration analysis.
  mm
    Anterior: number analyzed (Participants) | 344
    Anterior | 24.940 (4.811)
    Middle: number analyzed (Participants) | 344
    Middle | 24.207 (4.264)
    Posterior: number analyzed (Participants) | 344
    Posterior | 26.502 (4.397)

OUTCOME MEASURES:

1. Primary Outcome: Back Pain Change From Baseline at 3 Months
Description: Back pain was measured using NRS. Patients rated their back pain on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be."
Time Frame: Baseline, 3 months after surgery
Population: The number analyzed was based on the observed data and there were missing data stemming mostly from subject drop-out or lost-to-follow-ups. To some extent missing data were from unanswered questions, missing image, etc.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 350
units on a scale
  Back pain at baseline | 8.7 (1.2)
  Back pain at 3 Months: number analyzed (Participants) | 293
  Back pain at 3 Months | 2.7 (2.7)
  Back pain change: number analyzed (Participants) | 293
  Back pain change | -6.0 (3.0)

2. Primary Outcome: Back Function Change From Baseline by Oswestry Disability Index at 3 Months
Description: ODI Questionnaire was used to assess patient back function. The ODI score ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability).
Time Frame: Baseline, 3 months after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 350
units on a scale
  ODI score at baseline | 63.4 (14.9)
  ODI score at 3 months: number analyzed (Participants) | 283
  ODI score at 3 months | 27.1 (18.8)
  ODI change: number analyzed (Participants) | 283
  ODI change | -35.3 (20.5)

3. Primary Outcome: SF-36v2 Physical Component Summary Change From Baseline at 3 Months
Description: Quality of life was assessed by Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) version 2.0. The SF-36 v2 physical component summary (PCS) score is between 0 and 100, with higher scores denoting better quality of life.
Time Frame: Baseline, 3 months after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 346
units on a scale
  SF-36 PCS at baseline | 24.2 (7.0)
  SF-36 PCS at 3 months: number analyzed (Participants) | 279
  SF-36 PCS at 3 months | 36.6 (11.2)
  SF-36 PCS change: number analyzed (Participants) | 276
  SF-36 PCS change | 12.4 (11.4)

4. Primary Outcome: Change From Baseline in Quality of Life by the EQ-5D Index at 3 Months
Description: EQ-5D index scores range from 0 to 1.0 on a scale where 0 = death and 1.0 = perfect health.
Time Frame: Baseline, 3 months after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 348
units on a scale
  EQ-5D index at baseline | 0.383 (0.212)
  EQ-5D index at 3 months: number analyzed (Participants) | 281
  EQ-5D index at 3 months | 0.746 (0.194)
  EQ-5D index score change: number analyzed (Participants) | 279
  EQ-5D index score change | 0.351 (0.267)

5. Secondary Outcome: Back Pain
Description: as for outcome 1
Time Frame: Baseline, 7 days, 30 days, 6 months, 9 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 350
units on a scale
  Back pain at baseline | 8.7 (1.2)
  Back pain at 7 days: number analyzed (Participants) | 340
  Back pain at 7 days | 3.4 (2.3)
  Back pain at 30 days: number analyzed (Participants) | 315
  Back pain at 30 days | 3.2 (2.7)
  Back pain at 6 months: number analyzed (Participants) | 265
  Back pain at 6 months | 2.5 (2.7)
  Back pain at 9 months: number analyzed (Participants) | 277
  Back pain at 9 months | 2.3 (2.6)
  Back pain at 12 months: number analyzed (Participants) | 257
  Back pain at 12 months | 2.4 (2.8)

6. Secondary Outcome: Back Function (ODI)
Description: as for outcome 2
Time Frame: Baseline, 30 days, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 350
units on a scale
  ODI score at baseline | 63.4 (14.9)
  ODI score at 30 days: number analyzed (Participants) | 304
  ODI score at 30 days | 32.5 (19.5)
  ODI score at 6 months: number analyzed (Participants) | 255
  ODI score at 6 months | 25.7 (19.0)
  ODI score at 12 months: number analyzed (Participants) | 247
  ODI score at 12 months | 25.8 (19.0)

7. Secondary Outcome: Quality of Life by SF-36v2 PCS
Description: as for outcome 3
Time Frame: Baseline, 30 days, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 346
units on a scale
  SF-36 PCS at baseline | 24.2 (7.0)
  SF-36 PCS at 30 days: number analyzed (Participants) | 301
  SF-36 PCS at 30 days | 34.9 (9.8)
  SF-36 PCS at 6 months: number analyzed (Participants) | 253
  SF-36 PCS at 6 months | 37.6 (11.5)
  SF-36 PCS at 12 months: number analyzed (Participants) | 247
  SF-36 PCS at 12 months | 38.2 (12.1)

8. Secondary Outcome: Quality of Life by EQ-5D Index Score
Time Frame: Baseline, 30 days, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 348
units on a scale
  EQ-5D index at baseline | 0.383 (0.212)
  EQ-5D index at 30 days: number analyzed (Participants) | 302
  EQ-5D index at 30 days | 0.710 (0.196)
  EQ-5D index at 6 months: number analyzed (Participants) | 254
  EQ-5D index at 6 months | 0.756 (0.193)
  EQ-5D index at 12 months: number analyzed (Participants) | 245
  EQ-5D index at 12 months | 0.758 (0.193)

9. Secondary Outcome: Percentage of Subjects Having Daily Living Activities Limited Due to Back Pain in the Previous 2 Weeks
Time Frame: Baseline, 30 days, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 350
percentage of participants
  Baseline | 96.3
  30 days: number analyzed (Participants) | 304
  30 days | 53.3
  3 months: number analyzed (Participants) | 283
  3 months | 31.8
  6 months: number analyzed (Participants) | 255
  6 months | 31.0
  12 months: number analyzed (Participants) | 246
  12 months | 28.9

10. Secondary Outcome: The Number of Days With Limited Activities and Bed Rest Due to Back Pain in the Previous 2 Weeks;
Time Frame: Baseline, 30 days, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 350
days
  days of limited activities at baseline: number analyzed (Participants) | 349
  days of limited activities at baseline | 11.0 (4.6)
  days of bed rest at baseline: number analyzed (Participants) | 348
  days of bed rest at baseline | 6.0 (5.9)
  days of limited activities at 30 days: number analyzed (Participants) | 303
  days of limited activities at 30 days | 4.7 (5.7)
  days of bed rest at 30 days: number analyzed (Participants) | 304
  days of bed rest at 30 days | 1.5 (3.5)
  days of limited activities at 3 months: number analyzed (Participants) | 278
  days of limited activities at 3 months | 2.6 (4.6)
  days of bed rest at 3 months: number analyzed (Participants) | 280
  days of bed rest at 3 months | 0.7 (2.3)
  days of limited activities at 6 months: number analyzed (Participants) | 252
  days of limited activities at 6 months | 2.6 (4.8)
  days of bed rest at 6 months: number analyzed (Participants) | 253
  days of bed rest at 6 months | 0.7 (2.5)
  days of limited activities at 12 months: number analyzed (Participants) | 244
  days of limited activities at 12 months | 2.2 (4.5)
  days of bed rest at 12 months: number analyzed (Participants) | 245
  days of bed rest at 12 months | 0.7 (2.4)

11. Secondary Outcome: Ambulatory Status
Time Frame: Baseline, 7 days, 30 days, 3 months, 6 months, 9 months, and 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 350
percentage of participants
  Able to walk at baseline | 42.3
  Walk with aid at baseline | 50.3
  Unable to walk at baseline | 7.4
  Able to walk at 7 days: number analyzed (Participants) | 339
  Able to walk at 7 days | 59.9
  Walk with aid at 7 days: number analyzed (Participants) | 339
  Walk with aid at 7 days | 38.3
  Unable to walk at 7 days: number analyzed (Participants) | 339
  Unable to walk at 7 days | 1.8
  Able to walk at 30 days: number analyzed (Participants) | 315
  Able to walk at 30 days | 62.5
  Walk with aid at 30 days: number analyzed (Participants) | 315
  Walk with aid at 30 days | 36.2
  Unable to walk at 30 days: number analyzed (Participants) | 315
  Unable to walk at 30 days | 1.3
  Able to walk at 3 months: number analyzed (Participants) | 293
  Able to walk at 3 months | 64.5
  Walk with aid at 3 months: number analyzed (Participants) | 293
  Walk with aid at 3 months | 34.1
  Unable to walk at 3 months: number analyzed (Participants) | 293
  Unable to walk at 3 months | 1.4
  Able to walk at 6 months: number analyzed (Participants) | 266
  Able to walk at 6 months | 62.4
  Walk with aid at 6 months: number analyzed (Participants) | 266
  Walk with aid at 6 months | 36.1
  Unable to walk at 6 months: number analyzed (Participants) | 266
  Unable to walk at 6 months | 1.5
  Able to walk at 9 months: number analyzed (Participants) | 278
  Able to walk at 9 months | 68.7
  Walk with aid at 9 months: number analyzed (Participants) | 278
  Walk with aid at 9 months | 30.9
  Unable to walk at 9 months: number analyzed (Participants) | 278
  Unable to walk at 9 months | 0.4
  Able to walk at 12 months: number analyzed (Participants) | 258
  Able to walk at 12 months | 63.2
  Walk with aid at 12months: number analyzed (Participants) | 258
  Walk with aid at 12months | 35.7
  Unable to walk at 12 months: number analyzed (Participants) | 258
  Unable to walk at 12 months | 1.2

12. Secondary Outcome: Barthel Index (Only for Subjects With Osteoporosis)
Description: For subjects with osteoporosis, the Barthel index was used for rating subject activities of daily living on a scale from 0 (maximum disability) to 20 (no disability).
Time Frame: Baseline, 30 days, 3 months 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 343
units on a scale
  Barthel index score at baseline | 16.2 (4.0)
  Barthel index score at 30 days: number analyzed (Participants) | 299
  Barthel index score at 30 days | 18.8 (2.1)
  Barthel index score at 3 months: number analyzed (Participants) | 280
  Barthel index score at 3 months | 19.1 (2.0)
  Barthel index score at 6 months: number analyzed (Participants) | 253
  Barthel index score at 6 months | 19.1 (1.8)
  Barthel index score at 12 months: number analyzed (Participants) | 244
  Barthel index score at 12 months | 19.1 (1.8)

13. Secondary Outcome: Karnofsky Performance Scale
Description: For subjects with cancer, the Karnofsky performance scale was used for rating subject activities of daily living.The Karnofsky performance scale rates a subject on an 11-step scale from 0 (dead) to 100 (normal, no complaints, no evidence of disease), and a score of 70 is a clinically meaningful threshold for self-care.
Time Frame: Baseline, 30 days, 3 months 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 7
units on a scale
  Karnofsky performance scale at baseline | 75.7 (21.5)
  Karnofsky performance scale at 30 days: number analyzed (Participants) | 5
  Karnofsky performance scale at 30 days | 88.0 (11.0)
  Karnofsky performance scale at 3 months: number analyzed (Participants) | 4
  Karnofsky performance scale at 3 months | 90.0 (14.1)
  Karnofsky performance scale at 6 months: number analyzed (Participants) | 4
  Karnofsky performance scale at 6 months | 85.0 (30.0)
  Karnofsky performance scale at 12 months: number analyzed (Participants) | 3
  Karnofsky performance scale at 12 months | 96.7 (5.8)

14. Secondary Outcome: Vertebral Body Height Restoration (Absolute Height Restored as Percent, AHRP)
Description: AHRP (Absolute height restored as percent) was the amount of height restored in the vertebral body expressed as a percent of estimated pre-fracture (EP) height. Measurements were assessed at anterior, medial, and posterior locations on the vertebral body.
Time Frame: Baseline, pre-discharge, 3 months, and 12 months
Population: A total of 490 treated levels in 344 subjects were included in vertebral body height restoration analysis. The number analyzed was based on the observed data and there were missing data stemming mostly from subject drop-out or lost-to-follow-ups. To some extent missing data were from unanswered questions, missing image, etc.
Measure: Mean (Standard Deviation); unit: percentage of pre-fracture height
Units Other Than Participants: Treated levels
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 344
Number analyzed (Treated levels) | 490
percentage of pre-fracture height
  Anterior height Loss from EP at baseline: number analyzed (Participants) | 312
  Anterior height Loss from EP at baseline: number analyzed (Treated levels) | 435
  Anterior height Loss from EP at baseline | -26.438 (22.008)
  Middle height loss from EP at baseline: number analyzed (Participants) | 312
  Middle height loss from EP at baseline: number analyzed (Treated levels) | 435
  Middle height loss from EP at baseline | -27.719 (20.861)
  Posterior height loss from EP at baseline: number analyzed (Participants) | 312
  Posterior height loss from EP at baseline: number analyzed (Treated levels) | 435
  Posterior height loss from EP at baseline | -8.228 (10.966)
  Anterior AHRP at pre-discharge: number analyzed (Participants) | 291
  Anterior AHRP at pre-discharge: number analyzed (Treated levels) | 407
  Anterior AHRP at pre-discharge | 3.897 (9.822)
  Middle AHRP at pre-discharge: number analyzed (Participants) | 291
  Middle AHRP at pre-discharge: number analyzed (Treated levels) | 407
  Middle AHRP at pre-discharge | 4.205 (9.783)
  Posterior AHRP at pre-discharge: number analyzed (Participants) | 291
  Posterior AHRP at pre-discharge: number analyzed (Treated levels) | 407
  Posterior AHRP at pre-discharge | 1.280 (7.280)
  Anterior AHRP at 3 months: number analyzed (Participants) | 249
  Anterior AHRP at 3 months: number analyzed (Treated levels) | 340
  Anterior AHRP at 3 months | 1.511 (10.426)
  Middle AHRP at 3 months: number analyzed (Participants) | 249
  Middle AHRP at 3 months: number analyzed (Treated levels) | 340
  Middle AHRP at 3 months | 2.223 (10.076)
  Posterior AHRP at 3 months: number analyzed (Participants) | 249
  Posterior AHRP at 3 months: number analyzed (Treated levels) | 340
  Posterior AHRP at 3 months | 0.101 (7.474)
  Anterior AHRP at 12 months: number analyzed (Participants) | 203
  Anterior AHRP at 12 months: number analyzed (Treated levels) | 273
  Anterior AHRP at 12 months | 1.308 (10.765)
  Middle AHRP at 12 months: number analyzed (Participants) | 203
  Middle AHRP at 12 months: number analyzed (Treated levels) | 273
  Middle AHRP at 12 months | 1.567 (10.453)
  Posterior AHRP at 12 months: number analyzed (Participants) | 203
  Posterior AHRP at 12 months: number analyzed (Treated levels) | 273
  Posterior AHRP at 12 months | -0.028 (8.284)

15. Secondary Outcome: Vertebral Body Angle
Description: The vertebral body kyphosis angle (VBA) was defined as the angle formed by lines drawn parallel to the caudal and cranial fractured vertebral body endplates.
Time Frame: Baseline, pre-discharge, 3 months, and 12 months
Population: A total of 490 treated levels in 344 subjects were included in VBA analysis. The number analyzed was based on the observed data and there were missing data stemming mostly from subject drop-out or lost-to-follow-ups. To some extent missing data were from unanswered questions, missing image, etc.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Treated levels
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 344
Number analyzed (Treated levels) | 490
degrees
  vertebral body angle at baseline: number analyzed (Participants) | 313
  vertebral body angle at baseline: number analyzed (Treated levels) | 440
  vertebral body angle at baseline | -10.474 (8.152)
  Vertebral body angle at pre-discharge: number analyzed (Participants) | 317
  Vertebral body angle at pre-discharge: number analyzed (Treated levels) | 449
  Vertebral body angle at pre-discharge | -9.522 (6.867)
  Angle change from baseline at pre-discharge: number analyzed (Participants) | 291
  Angle change from baseline at pre-discharge: number analyzed (Treated levels) | 408
  Angle change from baseline at pre-discharge | 1.117 (4.137)
  Vertebral body angle at 3 months: number analyzed (Participants) | 269
  Vertebral body angle at 3 months: number analyzed (Treated levels) | 372
  Vertebral body angle at 3 months | -10.119 (6.781)
  Angle change from baseline at 3 months: number analyzed (Participants) | 249
  Angle change from baseline at 3 months: number analyzed (Treated levels) | 341
  Angle change from baseline at 3 months | 0.633 (4.282)
  Vertebral body angle at 12 months: number analyzed (Participants) | 227
  Vertebral body angle at 12 months: number analyzed (Treated levels) | 311
  Vertebral body angle at 12 months | -9.876 (6.714)
  Angle change from baseline at 12 months: number analyzed (Participants) | 204
  Angle change from baseline at 12 months: number analyzed (Treated levels) | 277
  Angle change from baseline at 12 months | 0.748 (4.315)

16. Secondary Outcome: Local Cobb Angle
Description: The local Cobb angle (LCA) was defined as the angle formed by lines drawn parallel to the superior endplate of the vertebral body above and the inferior endplate of the vertebral body below.
Time Frame: Baseline, pre-discharge, 3 months, and 12 months
Population: A total of 490 treated levels in 344 subjects were included in LCA analysis. The number analyzed was based on the observed data and there were missing data stemming mostly from subject drop-out or lost-to-follow-ups. To some extent missing data were from unanswered questions, missing image, etc.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Treated levels
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 344
Number analyzed (Treated levels) | 490
degrees
  Local Cobb angle at baseline: number analyzed (Participants) | 306
  Local Cobb angle at baseline: number analyzed (Treated levels) | 417
  Local Cobb angle at baseline | -12.919 (18.302)
  Local Cobb angle at pre-discharge: number analyzed (Participants) | 311
  Local Cobb angle at pre-discharge: number analyzed (Treated levels) | 429
  Local Cobb angle at pre-discharge | -11.190 (17.244)
  Angle change from baseline at pre-discharge: number analyzed (Participants) | 283
  Angle change from baseline at pre-discharge: number analyzed (Treated levels) | 382
  Angle change from baseline at pre-discharge | 2.707 (5.102)
  Local Cobb angle at 3 months: number analyzed (Participants) | 264
  Local Cobb angle at 3 months: number analyzed (Treated levels) | 359
  Local Cobb angle at 3 months | -13.439 (17.843)
  Angle change from baseline at 3 months: number analyzed (Participants) | 243
  Angle change from baseline at 3 months: number analyzed (Treated levels) | 322
  Angle change from baseline at 3 months | 0.253 (5.979)
  Local Cobb angle at 12 months: number analyzed (Participants) | 222
  Local Cobb angle at 12 months: number analyzed (Treated levels) | 299
  Local Cobb angle at 12 months | -12.819 (18.643)
  Angle change from baseline at 12 months: number analyzed (Participants) | 201
  Angle change from baseline at 12 months: number analyzed (Treated levels) | 264
  Angle change from baseline at 12 months | -0.197 (6.106)

17. Secondary Outcome: Subsequent Radiographic Fractures
Description: A subsequent VCF was defined as any fracture at an index or non-index vertebral body occurring after the initial procedure as compared to baseline. The percentage of subjects having one or more subsequent VCFs is presented.
Time Frame: 3 months and 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 267
percentage of participants
  Subsequent fractures at 3 months | 36.7
  Subsequent fractures at 12 months: number analyzed (Participants) | 246
  Subsequent fractures at 12 months | 47.6

18. Secondary Outcome: Neurological Success Rate
Description: Neurological functions were assessed preoperatively and postoperatively. Each of the individual functions was comprised of a number of elements. Investigators evaluated whether observations in each function category was normal or abnormal, and documentation of abnormal findings were required for each element in that function. Success for each component was defined as maintenance or improvement from preoperative for all elements. Success for overall neurologic status was defined as successful in all components.
Time Frame: Pre-discharge, 30 days, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty
Number analyzed (Participants) | 350
percentage of participants
  Neurological success at predischarge: number analyzed (Participants) | 337
  Neurological success at predischarge | 79.2
  Neurological success at 30 days: number analyzed (Participants) | 313
  Neurological success at 30 days | 76.7
  Neurological success at 3 months: number analyzed (Participants) | 292
  Neurological success at 3 months | 76.4
  Neurological success at 6 months: number analyzed (Participants) | 265
  Neurological success at 6 months | 74.3
  Neurological success at 12 months: number analyzed (Participants) | 257
  Neurological success at 12 months | 76.7

ADVERSE EVENTS:
Time Frame: Overall study about 12-month follow up
Arm/Group | Balloon Kyphoplasty
Serious Adverse Events (participants affected / at risk) | 79/350
Other Adverse Events (participants affected / at risk) | 128/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Kyphoplasty (N=350)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1)
Lupus hepatitis (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (3)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 11 (14)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (26)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Vascular stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Kyphoplasty (N=350)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrioventricular block (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Coeliac disease (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Device breakage (General disorders) | 1 (1)
Device malfunction (General disorders) | 1 (1)
Implant site extravasation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 9 (9)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 18 (18)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 4 (4)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (30)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 4 (5)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 10 (10)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 6 (6)
Scoliosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 4 (4)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 2 (2)
Spinal cord compression (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Labile hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less